CLINICAL TRIAL: NCT05414448
Title: Combination of Artificial Intelligence (ENDOAID) and Mucosal Exposure Device (ENDOCUFF) to Enhance Colorectal Neoplasia Detection: a Randomized Controlled Trial
Brief Title: Combination of Artificial Intelligence and Mucosal Exposure Device to Enhance Colorectal Neoplasia Detection
Acronym: AIDEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University Hospital Augsburg (Other); Changi General Hospital (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CREC2022.152
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Adenoma; Colorectal Cancer; Colorectal Neoplasms
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENDOAID (No Intervention): CADe system will be used during withdrawal phase of colonoscopy.
- ENDOAID with ENDOCUFF (Experimental): CADe system and mucosal exposure device (ENDOCUFF) will be used during withdrawal phase of colonoscopy.
  Interventions: Device: ENDOCUFF

INTERVENTIONS:
Device: ENDOCUFF — ENDOCUFF mucousal exposure device will be used during withdrawal process of the colonoscopy.
  Arms: ENDOAID with ENDOCUFF

SUMMARY:
The investigators hypothesize that the combined use of CADe system (ENDOAID) and mucosal exposure device (Endocuff Vision®) would improve the adenoma detection rate when compared to CADe system alone.

DETAILED DESCRIPTION:
High polyp miss rates were reported in standard colonoscopies. As a result, a significant proportion of interval CRC was attributed to the missed lesions during index colonoscopy. Risk factors of missed lesions included proximal location, serrate or flat morphology, poor bowel preparation, short withdrawal time and endoscopist experience.

To overcome this pitfall, various methods were developed to improve adenoma detection rate (ADR), including distal attachment devices. Among the mucosal exposure devices, Endocuff Vision® was shown to be superior than conventional colonoscopies.

Recently, artificial intelligence and automatic computer-aided polyp detection (CADe) systems have developed rapidly and revolutionized the medical field. Nevertheless, there was a potential limitation of 'blind spot' if the endoscopist failed to expose the colonic mucosa adequately leading to missed lesions. To date, no available data or ongoing clinical trial was reported regarding the combined use of CADe and mucosal exposure devices. It may enhance the performance of CADe and provide a novel definitive solution to this unaddressed yet important clinical problem.

In this prospective parallel randomized controlled trial, we aim to evaluate the impact of combined use of a new CADe system (ENDOAID) and mucosal exposure device (Endocuff Vision®) on colorectal neoplasia detection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 45-85 years old;
2. They require elective colonoscopy for colorectal cancer screening, polyp surveillance, or investigation of symptoms such as anemia or altered bowel habit;
3. Written informed consent obtained.

Exclusion Criteria:

1. Contraindication to colonoscopy (e.g. intestinal obstruction or perforation)
2. Contraindication or conditions precluding polyp resection (e.g. active gastrointestinal bleeding, uninterrupted anticoagulation or dual antiplatelets)
3. Staged procedure for polypectomy or biopsy of known unresected lesions
4. Previous surgical resection of colon
5. Personal history of colorectal cancer
6. Personal history of familial polyposis syndrome
7. Personal history of inflammatory bowel disease
8. Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above)
9. Pregnancy
10. Unable to obtain informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1726 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ADR | During the colonoscopy
  adenoma detection rate

SECONDARY OUTCOMES:
ADR for adenomas of different sizes | During the colonoscopy
  <5mm, 5-10mm, >10mm
ADR for adenomas of different colonic segments | During the colonoscopy
  caecum, ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid colon, rectum
Mean number of adenomas per colonoscopy | During the colonoscopy
  Mean number of adenomas per colonoscopy
Advanced adenoma detection rate | During the colonoscopy
  Advanced adenoma detection rate
Sessile serrated lesion (SSL) detection rate | During the colonoscopy
  Sessile serrated lesion (SSL) detection rate
Polyp detection rate | During the colonoscopy
  Polyp detection rate
Non-neoplastic resection rate | During the colonoscopy
  defined as absence of adenoma or SSL or cancer within resected specimen
Caecal intubation time | During the colonoscopy
  Caecal intubation time
Withdrawal time | During the colonoscopy
  excluding interventions
Total procedural time | During the colonoscopy
  Total procedural time
False positive rate | During the colonoscopy
  defined as computer artifacts due to colonic mucosal wall or bowel content lasting for >2 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: No